CLINICAL TRIAL: NCT01199692
Title: Characterization of Metabolic Biomarkers in Subjects of Varying Age, Gender, Ethnicity, Body Mass Distribution, Dietary Habits, Exercise Habits, Medication Requirements, and Disease State Burden
Brief Title: Characterization of Metabolic Biomarkers in Varying Subjects
Status: Completed | Type: Observational
Sponsor: CPL Associates (Other)
Responsible Party: Principal Investigator, Scott Monte, Program Director, CPL Associates
Other Study IDs: CPL201006A
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Age
- Gender
- Ethnicity
- Body Mass Distribution
- Dietary Habits
- Exercise Habits
- Medication Requirements
- Disease State Burden

SUMMARY:
Traditional dietary, lifestyle, behavioral and pharmacologic treatment strategies have proven relatively ineffective for treating obesity, and once metabolic abnormalities such as Type 2 Diabetes (T2D) develop, definitive strategies to prevent major cardiovascular events remain elusive. More positively, the identification of a scientific resolution for obesity and T2D in the short-term is not outside the bounds of reality. Because the complexity of metabolic regulation is likely to include already characterized biomarkers, as well as other unidentified factors, it is logical to sample subjects of various ages, gender, ethnicity, body mass distribution, dietary habits, exercise habits, medication requirements, and disease states to discover associations and pathways related to the restoration of normal metabolism.

DETAILED DESCRIPTION:
As an observational study design, study investigators will prospectively identify potential subjects from various primary care and/or specialty care clinics in Western New York. Prior to the commencement of any study procedures, subjects will document informed consent and acknowledgement of HIPPA rights. Following approval from their practitioner, subjects may be asked on multiple occasions to complete or undergo any or all of the following types of study procedures:

* Medical record review and follow-up
* Fasting blood sample (volume limitations stipulated within)
* Pre-meal, during meal, and post-meal blood sample (volume limits within)
* Short-term and/or long-term dietary intervention (MD approved)
* Short-term and/or long-term exercise intervention (MD approved)
* Blood glucose log
* Food and exercise diaries
* Pre- and post-medication blood sampling (neutraceutical or Rx products)
* 24-hour urine sampling
* Spot urine sampling
* Stool microbiologic sampling
* Intestinal microbiologic sampling (gastric bypass subjects only)

ELIGIBILITY:
Inclusion Criteria:

* Age =>18
* Weight =>110 pounds

Exclusion Criteria:

* Age <18
* Weight <110 pounds
* Pregnant
* Poor venous access or poor likelihood to adhere with study procedures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects of varying age, gender, ethnicity, body mass distribution, dietary habits, exercise habits, medication requirements and disease state burdens
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-08; Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Monte, PharmD, Principal Investigator — CPL Associates, LLC
Locations (1):
- Synergy Bariatrics, A Department of ECMC, Williamsville, New York, United States